CLINICAL TRIAL: NCT02059486
Title: Impact Evaluation of the Teen Choice Program
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Mathematica Policy Research, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PRP699104
Record Dates: First submitted 2014-01-30; First posted 2014-02-11 (Estimated); Last update posted 2017-04-17 (Actual); Status verified 2017-04

CONDITIONS: Sexual Behavior
MeSH Terms: conditions — Sexual Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Teen Choice (Experimental): The curriculum provides comprehensive sexual education on topics such as anatomy, puberty, sexually transmitted infections, and contraceptive methods (including abstinence). It also covers topics such as gender and sex roles, sexual orientation, decision making and conflict resolution, adult-teen relationships, rape and sexual assault, and coping with stress. The curriculum can be delivered in different formats that range in length from 6 to 12 weeks.
  Interventions: Behavioral: Teen Choice
- Control (No Intervention): Business as usual school health curriuclum

INTERVENTIONS:
Behavioral: Teen Choice — The curriculum provides sexual education on topics such as anatomy, puberty, sexually transmitted infections, and contraceptive methods (including abstinence). It also covers topics such as gender and sex roles, sexual orientation, decision making and conflict resolution, adult-teen relationships, rape and sexual assault, and coping with stress.
  Arms: Teen Choice

SUMMARY:
The purpose of this study is to evaluate the impact of the Teen Choice program on reducing the rates of unprotected sex of high risk youth in New York.

DETAILED DESCRIPTION:
This study uses a randomized controlled design to compare the impacts of the Teen Choice Program to the "business-as-usual" school curriculum. The Teen Choice curriculum is designed for adolescents aged 12 to 19 and will be delivered in different formats that range in length from 6 to 12 weeks. Teen Choice will be offered during the regular school day to middle and high school aged youth. This study is being conducted as part of the national Personal Responsibility Education Program evaluation funded by Administration for Children and Families within the U.S. Department of Health and Human Services.

ELIGIBILITY:
Inclusion Criteria:

* Age 12-19
* Attending one of the participating schools

Exclusion Criteria:

* Juvenile Justice Youth
* School clinician determined trauma histories
* School clinician determined developmental issues

Ages: 12 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 465 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2018-06 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Unprotected sex in the three months prior to the survey | 6-months post random assignment

SECONDARY OUTCOMES:
Sexual Initiation | 6-months post intervention

CONTACTS AND LOCATIONS:
Overall Officials: Robert Wood, PhD, Study Director — Mathematica Policy Research
Locations (5):
- United States (5):
  - R.O.A.D.S., Brooklyn, New York
  - Clark Academy, Dobbs Ferry, New York
  - Robert H Goddard High School, New York, New York
  - Bronx Community High School, The Bronx, New York
  - Biondi School, Yonkers, New York